CLINICAL TRIAL: NCT01568112
Title: A Randomized, Double-Blind, Phase 3b Study to Evaluate Effects of Aspirin or Dose Titration on Flushing and Gastrointestinal Events Following Oral Administration of BG00012 Dosed at 240 mg BID
Brief Title: Effect of Aspirin Pretreatment or Slow Dose Titration on Flushing and Gastrointestinal Events in Healthy Volunteers Receiving Delayed-release Dimethyl Fumarate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 109HV321
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Results first posted 2016-06-13 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: BG00012; gastrointestinal events; flushing events; dose titration; pre-medication; aspirin
MeSH Terms: interventions — Dimethyl Fumarate; Fumarates; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- BG00012 (Experimental): Participants received BG00012 for 8 weeks (120 mg BID during the first week and 240 mg BID during the subsequent 7 weeks) and premedication with ASA placebo during the first 4 weeks.
  Interventions: Drug: BG00012 (dimethyl fumarate); Drug: BG00012 placebo; Drug: ASA placebo
- Placebo (Placebo Comparator): Participants received BG00012 placebo for 8 weeks and premedication with ASA placebo during the first 4 weeks.
  Interventions: Drug: BG00012 placebo; Drug: ASA placebo
- BG00012 + ASA (Experimental): Participants received BG00012 for 8 weeks (120 mg BID during the first week and 240 mg BID during the subsequent 7 weeks) and premedication with ASA during the first 4 weeks.
  Interventions: Drug: BG00012 (dimethyl fumarate); Drug: BG00012 placebo; Drug: ASA
- BG00012 Slow Titration (Experimental): Participants received BG00012 for 8 weeks (120 mg once daily [QD] during Week 1, 120 mg BID during Week 2, 240 mg AM/120mg PM during Week 3, and 240 mg BID during Week 4, and 240 mg BID during Weeks 5 to 8) and premedication with ASA placebo during the first 4 weeks.
  Interventions: Drug: BG00012 (dimethyl fumarate); Drug: BG00012 placebo; Drug: ASA placebo

INTERVENTIONS:
Drug: BG00012 (dimethyl fumarate) — Each capsule contains 120 mg dimethyl fumarate (DMF). Fast titration involves taking one 120 mg capsule in the morning and one in the evening (240 mg daily) for one week, and then escalating to a dose of 480 mg daily (two capsules morning and evening) for the remainder of the study.Slow titration expands the dose escalation time to 4 weeks.
  Other Names: BG-12; oral fumarate; DMF
  Arms: BG00012; BG00012 + ASA; BG00012 Slow Titration
Drug: BG00012 placebo — Placebo matching BG00012
Drug: ASA — 325 mg microcoated aspirin (ASA)
  Other Names: acetylsalicylic acid; aspirin
  Arms: BG00012 + ASA
Drug: ASA placebo — Placebo matching aspirin
  Arms: BG00012; BG00012 Slow Titration; Placebo

SUMMARY:
The primary objective of the study is to evaluate whether premedication with 325 mg microcoated aspirin (ASA) tablet or a slow-titration dosing schedule of BG00012 reduces the incidence and severity of flushing and GI events following oral administration of BG00012 dosed at 240 mg twice a day (BID) in healthy volunteers. The secondary objective of this study is to evaluate the safety and tolerability of BG00012 when administered orally as a 240 mg BID dose regimen with and without 325 mg ASA premedication or following a slow-titration dosing schedule in healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

* Must give written informed consent and any authorizations required by local law
* Must have a body mass index (BMI) of between 18.0 to 34.0 kg/m^2,inclusive.
* Ability to complete the tolerability scales by accurately using the hand-held subject reporting device
* Subjects of childbearing potential must be willing to practice effective contraception

Key Exclusion Criteria:

* History of clinically significant diseases
* History of severe allergic or anaphylactic reactions
* Intolerance to aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs)
* Diarrhea, constipation, abdominal pain, flushing or nausea within 28 days prior to Day 1

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Saint Paul, Minnesota, United States

REFERENCES:
- [Result] O'Gorman J, Russell HK, Li J, Phillips G, Kurukulasuriya NC, Viglietta V. Effect of Aspirin Pretreatment or Slow Dose Titration on Flushing and Gastrointestinal Events in Healthy Volunteers Receiving Delayed-release Dimethyl Fumarate. Clin Ther. 2015 Jul 1;37(7):1402-1419.e5. doi: 10.1016/j.clinthera.2015.03.028. Epub 2015 May 19. PMID 25999183

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Started | 44 | 44 | 43 | 42
Completed | 39 | 36 | 36 | 30
Not Completed | 5 | 8 | 7 | 12
Not completed — Randomized But Not Treated | 0 | 1 | 0 | 0
Not completed — Withdrew due to Adverse Event | 2 | 4 | 6 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 7
Not completed — Withdrawal by Physician | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized and treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration | Total
Number analyzed (Participants) | 44 | 43 | 43 | 42 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (8.78) | 39.0 (9.61) | 38.1 (10.29) | 36.2 (9.33) | 37.2 (9.54)
Age, Customized [Number; unit: participants]
  25 to 34 years | 22 | 19 | 17 | 21 | 79
  35 to 44 years | 13 | 7 | 13 | 10 | 43
  45 to 55 years | 9 | 17 | 13 | 11 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 21 | 17 | 20 | 72
  Male | 30 | 22 | 26 | 22 | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Overall Flushing Events During the Overall Treatment Period, as Assessed by the Modified Flushing Severity Scale (MFSS)
Description: Participant-reported flushing side effect events during the treatment period recorded on the eDiary as assessed by MFSS. MFSS questionnaire measures the side effects related to flushing following drug administration. Flushing means redness, warmth, tingling or itching of the skin. This questionnaire relates only to the period of time since the investigational drug was administered and was to be completed within 10 hours of taking the study drug (2 times/day). Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects).
Time Frame: Day 1 to Week 8
Population: Participants who received at least 1 dose of study medication and who had at least 1 diary entry of the relevant questionnaire data during the visit interval.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 43 | 42
percentage of participants
  Overall flushing events | 41 | 91 | 81 | 98
  Overall redness events | 27 | 86 | 77 | 90
  Overall warmth events | 41 | 93 | 84 | 98
  Overall tingling events | 23 | 88 | 67 | 86
  Overall itching events | 20 | 86 | 72 | 98
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Overall flushing events; Test type: Superiority or Other; Difference in percentage = -9, 95% CI 2-sided [-30.8 to 12.9] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Overall flushing events; Test type: Superiority or Other; Difference in percentage = 7, 95% CI 2-sided [-14.1 to 27.8] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 3: Comparison: BG00012 vs BG00012 + ASA; Overall redness events; Test type: Superiority or Other; Difference in percentage = -9, 95% CI 2-sided [-30.8 to 12.9] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 4: Comparison: BG00012 vs BG00012 Slow Titration; Overall redness events; Test type: Superiority or Other; Difference in percentage = 4, 95% CI 2-sided [-16.4 to 25.5] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 5: Comparison: BG00012 vs BG00012 + ASA; Overall tingling events; Test type: Superiority or Other; Difference in percentage = -21, 95% CI 2-sided [-41.7 to 1.3] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 6: Comparison: BG00012 vs BG00012 Slow Titration; Overall tingling events; Test type: Superiority or Other; Difference in percentage = -3, 95% CI 2-sided [-23.3 to 18.7] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 7: Comparison: BG00012 vs BG00012 + ASA; Overall itching events; Test type: Superiority or Other; Difference in percentage = -14, 95% CI 2-sided [-35.2 to 8.3] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 8: Comparison: BG00012 vs BG00012 Slow Titration; Overall itching events; Test type: Superiority or Other; Difference in percentage = 12, 95% CI 2-sided [-9.5 to 32.2] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 9: Comparison: BG00012 vs BG00012 + ASA; Overall warmth events; Test type: Superiority or Other; Difference in percentage = -9, 95% CI 2-sided [-30.8 to 12.9] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 10: Comparison: BG00012 vs BG00012 Slow Titration; Overall warmth events; Test type: Superiority or Other; Difference in percentage = 5, 95% CI 2-sided [-16.4 to 25.5] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

2. Primary Outcome: Percentage of Participants Reporting Overall Flushing Events During Weeks 1 to 4 (Combined), as Assessed by MFSS
Description: Participant-reported flushing side effect events during Weeks 1 to 4 recorded on the eDiary as assessed by MFSS. MFSS questionnaire measures the side effects related to flushing following drug administration. Flushing means redness, warmth, tingling or itching of the skin. This questionnaire relates only to the period of time since the investigational drug was administered and was to be completed within 10 hours of taking the study drug (2 times/day). Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects).
Time Frame: Week 1 to Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- BG00012 Slow Titration: Participants received BG00012 for 8 weeks (120 mg QD during Week 1, 120 mg BID during Week 2, 240 mg AM/120mg PM during Week 3, and 240 mg BID during Week 4, and 240 mg BID during Weeks 5 to 8) and premedication with ASA placebo during the first 4 weeks.
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 43 | 42
percentage of participants
  Overall flushing events | 41 | 86 | 72 | 98
  Overall redness events | 25 | 81 | 63 | 88
  Overall warmth events | 41 | 88 | 67 | 95
  Overall tingling events | 23 | 84 | 51 | 83
  Overall itching events | 16 | 77 | 56 | 95
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Overall flushing events; Test type: Superiority or Other; Difference in percentage = -14, 95% CI 2-sided [-35.2 to 8.3] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Overall flushing events; Test type: Superiority or Other; Difference in percentage = 12, 95% CI 2-sided [-9.5 to 32.2] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 3: Comparison: BG00012 vs BG00012 + ASA; Redness events; Test type: Superiority or Other; Difference in percentage = -19, 95% CI 2-sided [-39.6 to 3.7] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 4: Comparison: BG00012 vs BG00012 Slow Titration; Redness events; Test type: Superiority or Other; Difference in percentage = 7, 95% CI 2-sided [-14.1 to 27.8] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 5: Comparison: BG00012 vs BG00012 + ASA; Warmth events; Test type: Superiority or Other; Difference in percentage = -21, 95% CI 2-sided [-41.7 to 1.3] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 6: Comparison: BG00012 vs BG00012 Slow Titration; Warmth events; Test type: Superiority or Other; Difference in percentage = 7, 95% CI 2-sided [-14.1 to 27.8] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 7: Comparison: BG00012 vs BG00012 + ASA; Tingling events; Test type: Superiority or Other; Difference in percentage = -33, 95% CI 2-sided [-52.2 to -10.6] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 8: Comparison: BG00012 vs BG00012 Slow Titration; Tingling events; Test type: Superiority or Other; Difference in percentage = -0, 95% CI 2-sided [-21.0 to 21.0] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 9: Comparison: BG00012 vs BG00012 + ASA; Itching events; Test type: Superiority or Other; Difference in percentage = -21, 95% CI 2-sided [-41.7 to 1.3] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 10: Comparison: BG00012 vs BG00012 Slow Titration; Itching events; Test type: Superiority or Other; Difference in percentage = 18, 95% CI 2-sided [-2.4 to 38.8] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

3. Primary Outcome: Percentage of Participants Reporting Overall Flushing Events During Weeks 5 to 8 (Combined), as Assessed by MFSS
Description: as for outcome 2
Time Frame: Week 5 to Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 41 | 37 | 36 | 33
percentage of participants
  Overall flushing events | 24 | 86 | 72 | 85
  Overall redness events | 15 | 78 | 64 | 79
  Overall warmth events | 17 | 86 | 75 | 82
  Overall tingling events | 15 | 81 | 64 | 70
  Overall itching events | 22 | 78 | 58 | 61
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Overall flushing events; Test type: Superiority or Other; Difference in percentage = -14, 95% CI 2-sided [-35.6 to 9.2] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Overall flushing events; Test type: Superiority or Other; Difference in percentage = -2, 95% CI 2-sided [-24.7 to 21.7] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 3: Comparison: BG00012 vs BG00012 + ASA; Redness events; Test type: Superiority or Other; Difference in percentage = -14, 95% CI 2-sided [-35.6 to 9.2] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 4: Comparison: BG00012 vs BG00012 Slow Titration; Redness events; Test type: Superiority or Other; Difference in percentage = 0, 95% CI 2-sided [-22.9 to 23.7] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 5: Comparison: BG00012 vs BG00012 + ASA; Warmth events; Test type: Superiority or Other; Difference in percentage = -11, 95% CI 2-sided [-33.0 to 11.9] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 6: Comparison: BG00012 vs BG00012 Slow Titration; Warmth events; Test type: Superiority or Other; Difference in percentage = -5, 95% CI 2-sided [-27.5 to 18.8] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 7: Comparison: BG00012 vs BG00012 + ASA; Tingling events; Test type: Superiority or Other; Difference in percentage = -17, 95% CI 2-sided [-38.1 to 6.5] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 8: Comparison: BG00012 vs BG00012 Slow Titration; Tingling events; Test type: Superiority or Other; Difference in percentage = -11, 95% CI 2-sided [-34.2 to 12.2] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 9: Comparison: BG00012 vs BG00012 + ASA; Itching events; Test type: Superiority or Other; Difference in percentage = -20, 95% CI 2-sided [-40.6 to 3.8] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 10: Comparison: BG00012 vs BG00012 Slow Titration; Itching events; Test type: Superiority or Other; Difference in percentage = -18, 95% CI 2-sided [-40.2 to 5.5] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

4. Primary Outcome: Worst Severity Scores of Overall Flushing During Weeks 1 to 4 of Treatment (Combined), as Assessed by MFSS
Description: Worst severity of participant-reported flushing events during Weeks 1-4 of treatment combined, recorded on the eDiary as assessed by MFSS. MFSS questionnaire measures the side effects related to flushing following drug administration. Flushing means redness, warmth, tingling or itching of the skin. This questionnaire relates only to the period of time since the investigational drug was administered and was to be completed within 10 hours of taking the study drug (2 times/day). Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects).
Time Frame: Day 1 to Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 43 | 42
units on a scale
  Overall flushing | 1.2 (1.70) | 4.4 (2.68) | 2.4 (2.26) | 5.6 (2.24)
  Redness | 0.7 (1.33) | 3.8 (2.76) | 1.6 (1.75) | 5.1 (2.93)
  Warmth | 1.2 (1.76) | 4.0 (2.55) | 2.3 (2.17) | 5.2 (2.37)
  Tingling | 0.5 (1.00) | 3.4 (2.21) | 1.6 (2.13) | 4.0 (2.62)
  Itching | 0.5 (1.21) | 3.2 (2.45) | 1.3 (1.72) | 4.3 (2.10)
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Overall flushing events; Test type: Superiority or Other; Mean difference = -1.9, 95% CI 2-sided [-3.0 to -0.9], Standard Error of Mean 0.53 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Overall flushing events; Test type: Superiority or Other; Mean difference = 1.2, 95% CI 2-sided [0.2 to 2.3], Standard Error of Mean 0.54 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 3: Comparison: BG00012 vs BG00012 + ASA; Redness events; Test type: Superiority or Other; Mean difference = -2.2, 95% CI 2-sided [-3.2 to -1.2], Standard Error of Mean 0.50 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 4: Comparison: BG00012 + ASA vs BG00012 Slow Titration; Redness events; Test type: Superiority or Other; Mean difference = 1.3, 95% CI 2-sided [0.1 to 2.5], Standard Error of Mean 0.62 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 5: Comparison: BG00012 vs BG00012 + ASA; Warmth events; Test type: Superiority or Other; Mean difference = -1.7, 95% CI 2-sided [-2.8 to -0.7], Standard Error of Mean 0.51 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 6: Comparison: BG00012 + ASA vs BG00012 Slow Titration; Warmth events; Test type: Superiority or Other; Mean difference = 1.2, 95% CI 2-sided [0.1 to 2.3], Standard Error of Mean 0.53 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 7: Comparison: BG00012 vs BG00012 + ASA; Tingling events; Test type: Superiority or Other; Mean difference = -1.8, 95% CI 2-sided [-2.7 to -0.9], Standard Error of Mean 0.47 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 8: Comparison: BG00012 + ASA vs BG00012 Slow Titration; Tingling events; Test type: Superiority or Other; Mean difference = 0.6, 95% CI 2-sided [-0.4 to 1.6], Standard Error of Mean 0.52 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 9: Comparison: BG00012 vs BG00012 + ASA; Itching events; Test type: Superiority or Other; Mean difference = -1.9, 95% CI 2-sided [-2.8 to -1.0], Standard Error of Mean 0.46 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 10: Comparison: BG00012 + ASA vs BG00012 Slow Titration; Itching events; Test type: Superiority or Other; Mean difference = 1.2, 95% CI 2-sided [0.2 to 2.2], Standard Error of Mean 0.50 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

5. Primary Outcome: Worst Severity Scores of Overall Flushing During Weeks 5 to 8 of Treatment (Combined), as Assessed by MFSS
Description: Worst severity of participant-reported flushing events during Weeks 1-4 of treatment combined, recorded on the eDiary as assessed by MFSS. MFSS questionnaire measures the side effects related to flushing following drug administration. Flushing means redness, warmth, tingling or itching of the skin.This questionnaire relates only to the period of time since the investigational drug was administered and was to be completed within 10 hours of taking the study drug (2 times/day). Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects).
Time Frame: Week 5 to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 41 | 37 | 36 | 33
units on a scale
  Overall flushing | 0.9 (1.67) | 3.8 (2.48) | 3.3 (2.78) | 3.1 (2.26)
  Redness | 0.4 (1.14) | 3.6 (2.73) | 2.9 (2.67) | 2.9 (2.30)
  Warmth | 0.8 (1.79) | 3.9 (2.53) | 3.1 (2.50) | 2.9 (2.15)
  Tingling | 0.3 (0.82) | 3.3 (2.50) | 2.3 (2.36) | 2.2 (1.96)
  Itching | 0.7 (1.58) | 3.1 (2.71) | 2.3 (2.52) | 1.8 (2.04)
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Overall flushing events; Test type: Superiority or Other; Mean difference = -0.5, 95% CI 2-sided [-1.7 to 0.8], Standard Error of Mean 0.62 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Overall flushing events; Test type: Superiority or Other; Mean difference = -0.7, 95% CI 2-sided [-1.8 to 0.4], Standard Error of Mean 0.57 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 3: Comparison: BG00012 vs BG00012 + ASA; Redness events; Test type: Superiority or Other; Mean difference = -0.7, 95% CI 2-sided [-2.0 to 0.6], Standard Error of Mean 0.63 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 4: Comparison: BG00012 vs BG00012 Slow Titration; Redness events; Test type: Superiority or Other; Mean difference = -0.7, 95% CI 2-sided [-1.9 to 0.5], Standard Error of Mean 0.61 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 5: Comparison: BG00012 vs BG00012 + ASA; Warmth events; Test type: Superiority or Other; Mean difference = -0.8, 95% CI 2-sided [-2.0 to 0.4], Standard Error of Mean 0.59 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 6: Comparison: BG00012 vs BG00012 Slow Titration; Warmth events; Test type: Superiority or Other; Mean difference = -0.9, 95% CI 2-sided [-2.1 to 0.2], Standard Error of Mean 0.56 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 7: Comparison: BG00012 vs BG00012 + ASA; Tingling events; Test type: Superiority or Other; Mean difference = -1.0, 95% CI 2-sided [-2.2 to 0.1], Standard Error of Mean 0.57 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 8: Comparison: BG00012 vs BG00012 Slow Titration; Tingling events; Test type: Superiority or Other; Mean difference = -1.1, 95% CI 2-sided [-2.2 to -0.0], Standard Error of Mean 0.54 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 9: Comparison: BG00012 vs BG00012 + ASA; Itching events; Test type: Superiority or Other; Mean difference = -0.8, 95% CI 2-sided [-2.1 to 0.4], Standard Error of Mean 0.61 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 10: Comparison: BG00012 vs BG00012 Slow Titration; Itching events; Test type: Superiority or Other; Mean difference = -1.3, 95% CI 2-sided [-2.4 to -0.1], Standard Error of Mean 0.58 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

6. Primary Outcome: Percentage of Participants Reporting Overall Flushing Events During the Overall Treatment Period, as Assessed by the Modified Global Flushing Severity Scale (MGFSS)
Description: Participant-reported flushing events during the overall treatment period, recorded on the hand-held participant reporting device (eDiary) as assessed by MGFSS. The MGFSS measures the side effects related to flushing during the past 24 hours. Flushing means redness, warmth, tingling or itching of the skin. Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects). Day 1 data are not included in the analysis because MGFSS question refers to events reported in the 24 hours after the first dose on Day 1.
Time Frame: Day 2 to Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 42 | 42
percentage of participants | 43 | 86 | 74 | 93
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Overall flushing events; Test type: Superiority or Other; Difference in percentage = -12, 95% CI 2-sided [-32.2 to 9.5] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Overall flushing events; Test type: Superiority or Other; Difference in percentage = 7, 95% CI 2-sided [-14.1 to 27.8] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

7. Primary Outcome: Percentage of Participants Reporting Overall Flushing Events During Weeks 1 to 4 of Treatment (Combined), as Assessed by MGFSS
Description: Participant-reported flushing events during Weeks 1 to 4 of treatment (combined), recorded on the hand-held participant reporting device (eDiary) as assessed by MGFSS. The MGFSS measures the side effects related to flushing during the past 24 hours. Flushing means redness, warmth, tingling or itching of the skin. Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects). Day 1 data are not included in the analysis because MGFSS question refers to events reported in the 24 hours after the first dose on Day 1.
Time Frame: Day 2 to Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 42 | 42
percentage of participants | 41 | 84 | 62 | 90
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Test type: Superiority or Other; Difference in percentage = -22, 95% CI 2-sided [-41.0 to 0.1] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Test type: Superiority or Other; Difference in percentage = 7, 95% CI 2-sided [-14.1 to 27.8] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

8. Primary Outcome: Percentage of Participants Reporting Overall Flushing Events During Weeks 5 to 8 of Treatment (Combined), as Assessed by MGFSS
Description: Participant-reported flushing events during Weeks 5 to 8 of treatment (combined), recorded on the hand-held participant reporting device (eDiary) as assessed by MGFSS. The MGFSS measures the side effects related to flushing during the past 24 hours. Flushing means redness, warmth, tingling or itching of the skin. Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects). Day 1 data are not included in the analysis because MGFSS question refers to last 24 hours flushing score.
Time Frame: Week 5 to Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 41 | 37 | 36 | 33
percentage of participants | 24 | 86 | 67 | 85
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Test type: Superiority or Other; Difference in percentage = -20, 95% CI 2-sided [-40.6 to 3.8] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Test type: Superiority or Other; Difference in percentage = -2, 95% CI 2-sided [-24.7 to 21.7] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

9. Primary Outcome: Percentage of Participants Reporting Gastrointestinal (GI) Events During the Overall Treatment Period, as Assessed by the Modified Acute Gastrointestinal Scale (MAGISS)
Description: The MAGISS is a participant-reported questionnaire about side effects of the gastrointestinal system following drug administration, and is based on a 0- to 10-point scale, with 0 representing absence of symptoms and 10 representing the most severe symptoms. A participant was considered having overall GI side effect if he/she had a score of >=1 for at least one of the GI side effects including nausea, diarrhea, upper abdominal pain, lower abdominal pain, vomiting, indigestion, constipation, bloating and flatulence.
Time Frame: Day 1 to Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 43 | 42
percentage of participants | 73 | 81 | 81 | 86
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Test type: Superiority or Other; Difference in percentage = 0, 95% CI 2-sided [-22.0 to 22.0] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Test type: Superiority or Other; Difference in percentage = 4, 95% CI 2-sided [-16.4 to 25.5] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

10. Primary Outcome: Percentage of Participants Reporting GI Events During Weeks 1 to 4 of Treatment (Combined), as Assessed by MAGISS
Description: as for outcome 9
Time Frame: Day 1 to Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 43 | 42
percentage of participants | 66 | 81 | 79 | 79
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Test type: Superiority or Other; Difference in percentage = -2, 95% CI 2-sided [-24.2 to 19.7] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Test type: Superiority or Other; Difference in percentage = -3, 95% CI 2-sided [-23.3 to 18.7] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

11. Primary Outcome: Percentage of Participants Reporting GI Events During Weeks 5 to 8 of Treatment (Combined), as Assessed by MAGISS
Description: as for outcome 9
Time Frame: Week 5 to Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 41 | 37 | 36 | 33
percentage of participants | 41 | 59 | 53 | 61
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Test type: Superiority or Other; Difference in percentage = -7, 95% CI 2-sided [-29.4 to 17.1] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Test type: Superiority or Other; Difference in percentage = 1, 95% CI 2-sided [-22.1 to 24.5] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

12. Primary Outcome: Worst Severity Scores of Acute GI Events During Weeks 1 to 4 of Treatment (Combined), as Assessed by MAGISS
Description: Severity of GI-related events using the MAGISS to measure GI symptoms (nausea, diarrhea, upper abdominal pain, lower abdominal pain, vomiting, indigestion, constipation, bloating, flatulence), based on a 0- to 10-point scale, with 0 representing absence of symptoms and 10 representing the most severe symptoms.
Time Frame: Day 1 to Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 43 | 42
units on a scale
  Nausea | 0.7 (1.59) | 1.6 (2.41) | 1.6 (2.54) | 1.5 (2.09)
  Diarrhea | 1.0 (1.97) | 1.8 (2.47) | 1.5 (2.76) | 1.0 (1.67)
  Upper abdominal pain | 0.8 (1.38) | 1.1 (2.16) | 1.7 (2.71) | 1.4 (2.47)
  Lower abdominal pain | 0.5 (1.21) | 1.4 (2.14) | 1.3 (2.32) | 1.2 (2.12)
  Vomiting | 0.2 (0.75) | 0.3 (1.28) | 0.3 (1.63) | 0.2 (1.10)
  Indigestion | 0.7 (1.29) | 0.9 (1.83) | 0.6 (1.26) | 0.9 (1.97)
  Constipation | 0.4 (1.45) | 0.9 (2.23) | 0.6 (1.45) | 0.9 (1.85)
  Bloating | 0.5 (1.17) | 1.1 (1.96) | 1.3 (2.08) | 1.0 (1.88)
  Flatulence | 1.3 (1.73) | 1.3 (2.03) | 1.4 (1.76) | 1.6 (2.20)
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Nausea; Test type: Superiority or Other; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-1.1 to 1.1], Standard Error of Mean 0.53 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Nausea; Test type: Superiority or Other; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.1 to 0.9], Standard Error of Mean 0.49 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 3: Comparison: BG00012 vs BG00012 + ASA; Diarrhea; Test type: Superiority or Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.4 to 0.8], Standard Error of Mean 0.57 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 4: Comparison: BG00012 vs BG00012 Slow Titration; Diarrhea; Test type: Superiority or Other; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.7 to 0.1], Standard Error of Mean 0.46 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 5: Comparison: BG00012 vs BG00012 + ASA; Upper abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.5 to 1.6], Standard Error of Mean 0.53 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 6: Comparison: BG00012 vs BG00012 Slow Titration; Upper abdominal pain; Test type: Superiority or Other; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.7 to 1.3], Standard Error of Mean 0.50 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 7: Comparison: BG00012 vs BG00012 + ASA; Lower abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-1.0 to 0.9], Standard Error of Mean 0.48 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 8: Comparison: BG00012 vs BG00012 Slow Titration; Lower abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.1 to 0.8], Standard Error of Mean 0.46 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 9: Comparison: BG00012 vs BG00012 + ASA; Vomiting; Test type: Superiority or Other; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.6 to 0.7], Standard Error of Mean 0.32 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 10: Comparison: BG00012 vs BG00012 Slow Titration; Vomiting; Test type: Superiority or Other; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.6 to 0.5], Standard Error of Mean 0.26 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 11: Comparison: BG00012 vs BG00012 + ASA; Indigestion; Test type: Superiority or Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.0 to 0.3], Standard Error of Mean 0.34 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 12: Comparison: BG00012 vs BG00012 Slow Titration; Indigestion; Test type: Superiority or Other; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.8 to 0.8], Standard Error of Mean 0.41 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 13: Comparison: BG00012 vs BG00012 + ASA; Constipation; Test type: Superiority or Other; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.0 to 0.6], Standard Error of Mean 0.41 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 14: Comparison: BG00012 vs BG00012 Slow Titration; Constipation; Test type: Superiority or Other; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.8 to 0.9], Standard Error of Mean 0.44 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 15: Comparison: BG00012 vs BG00012 + ASA; Bloating; Test type: Superiority or Other; Difference in percentage = 0.2, 95% CI 2-sided [-0.7 to 1.1], Standard Error of Mean 0.4
Statistical Analysis 16: Comparison: BG00012 vs BG00012 Slow Titration; Bloating; Test type: Superiority or Other; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.9 to 0.7], Standard Error of Mean 0.42 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 17: Comparison: BG00012 vs BG00012 + ASA; Flatulence; Test type: Superiority or Other; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.8 to 0.9], Standard Error of Mean 0.41 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 18: Comparison: BG00012 vs BG00012 Slow Titration; Flatulence; Test type: Superiority or Other; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.7 to 1.1], Standard Error of Mean 0.46 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

13. Primary Outcome: Worst Severity Scores of Acute GI Events During Weeks 5 to 8 of Treatment (Combined), as Assessed by MAGISS
Description: as for outcome 12
Time Frame: Week 5 to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 41 | 37 | 36 | 33
units on a scale
  Nausea | 0.4 (1.51) | 0.9 (1.79) | 0.8 (1.94) | 0.9 (1.65)
  Diarrhea | 1.0 (2.01) | 1.4 (2.29) | 0.8 (2.13) | 0.7 (1.42)
  Upper abdominal pain | 0.6 (1.69) | 0.5 (1.50) | 0.4 (1.21) | 0.6 (1.56)
  Lower abdominal pain | 0.6 (1.48) | 0.4 (1.42) | 0.5 (1.38) | 0.9 (1.72)
  Vomiting | 0.2 (1.41) | 0.1 (0.82) | 0.1 (0.83) | 0.0 (0.00)
  Indigestion | 0.4 (1.26) | 0.5 (1.32) | 0.5 (1.38) | 0.4 (1.06)
  Constipation | 0.4 (1.20) | 0.1 (0.59) | 0.6 (1.63) | 0.3 (1.05)
  Bloating | 0.5 (1.23) | 0.7 (1.61) | 0.7 (1.55) | 0.8 (1.52)
  Flatulence | 0.8 (1.65) | 1.2 (2.04) | 0.4 (1.08) | 0.9 (1.54)
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Nausea; Test type: Superiority or Other; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.0 to 0.8], Standard Error of Mean 0.44 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Nausea; Test type: Superiority or Other; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.8 to 0.8], Standard Error of Mean 0.41 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 3: Comparison: BG00012 vs BG00012 + ASA; Diarrhea; Test type: Superiority or Other; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.7 to 0.4], Standard Error of Mean 0.52 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 4: Comparison: BG00012 vs BG00012 Slow Titration; Diarrhea; Test type: Superiority or Other; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.7 to 0.2], Standard Error of Mean 0.46 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 5: Comparison: BG00012 vs BG00012 + ASA; Upper abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.6], Standard Error of Mean 0.32 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 6: Comparison: BG00012 vs BG00012 Slow Titration; Upper abdominal pain; Test type: Superiority or Other; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.7 to 0.8], Standard Error of Mean 0.37 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 7: Comparison: BG00012 vs BG00012 + ASA; Lower abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.6 to 0.7], Standard Error of Mean 0.33 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 8: Comparison: BG00012 vs BG00012 Slow Titration; Lower abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.2 to 1.3], Standard Error of Mean 0.38 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 9: Comparison: BG00012 vs BG00012 + ASA; Vomiting; Test type: Superiority or Other; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.4], Standard Error of Mean 0.19 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 10: Comparison: BG00012 vs BG00012 Slow Titration; Vomiting; Test type: Superiority or Other; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.14 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 11: Comparison: BG00012 vs BG00012 + ASA; Indigestion; Test type: Superiority or Other; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.6 to 0.6], Standard Error of Mean 0.32 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 12: Comparison: BG00012 vs BG00012 Slow Titration; Indigestion; Test type: Superiority or Other; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.5], Standard Error of Mean 0.29 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 13: Comparison: BG00012 vs BG00012 + ASA; Constipation; Test type: Superiority or Other; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.1 to 1.0], Standard Error of Mean 0.28 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 14: Comparison: BG00012 vs BG00012 Slow Titration; Constipation; Test type: Superiority or Other; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.6], Standard Error of Mean 0.20 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 15: Comparison: BG00012 vs BG00012 + ASA; Bloating; Test type: Superiority or Other; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.8 to 0.7], Standard Error of Mean 0.37 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 16: Comparison: BG00012 vs BG00012 Slow Titration; Bloating; Test type: Superiority or Other; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.7 to 0.8], Standard Error of Mean 0.38 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 17: Comparison: BG00012 vs BG00012 + ASA; Flatulence; Test type: Superiority or Other; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.6 to -0.0], Standard Error of Mean 0.38 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 18: Comparison: BG00012 vs BG00012 Slow Titration; Flatulence; Test type: Superiority or Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.2 to 0.5], Standard Error of Mean 0.44 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

14. Primary Outcome: Percentage of Participants Reporting GI Events During the Overall Treatment Period, as Assessed by the Modified Overall Gastrointestinal Symptom Scale (MOGISS)
Description: The MOGISS is a questionnaire about overall side effects related to the gastrointestinal system (including nausea, diarrhea, upper abdominal pain, lower abdominal pain, vomiting, indigestion, constipation, bloating, and flatulence) during the 24 hours prior to each AM dose. Participants were to answer the questions at the same time each day, before the morning drug administration.
Time Frame: Day 1 to Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 42 | 42
percentage of participants | 59 | 70 | 79 | 79
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Test type: Superiority or Other; Difference in percentage = 9, 95% CI 2-sided [-11.8 to 30.0] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Test type: Superiority or Other; Difference in percentage = 9, 95% CI 2-sided [-11.8 to 30.0] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

15. Primary Outcome: Percentage of Participants Reporting GI Events During Weeks 1 to 4 (Combined), as Assessed by the Modified Overall Gastrointestinal Symptom Scale (MOGISS)
Description: as for outcome 14
Time Frame: Week 1 to Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 42 | 42
percentage of participants | 57 | 65 | 67 | 71
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Test type: Superiority or Other; Difference in percentage = 2, 95% CI 2-sided [-18.8 to 23.3] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Test type: Superiority or Other; Difference in percentage = 6, 95% CI 2-sided [-14.1 to 27.8] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

16. Primary Outcome: Percentage of Participants Reporting GI Events During Weeks 5 to 8 (Combined), as Assessed by the Modified Overall Gastrointestinal Symptom Scale (MOGISS)
Description: as for outcome 14
Time Frame: Week 5 to Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 41 | 37 | 36 | 33
percentage of participants | 34 | 59 | 50 | 58
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Test type: Superiority or Other; Difference in percentage = -9, 95% CI 2-sided [-32.1 to 14.3] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Test type: Superiority or Other; Difference in percentage = -2, 95% CI 2-sided [-25.0 to 21.7] — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

17. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious AEs (SAEs)
Description: AE: any untoward medical occurrence that does not necessarily have a causal relationship with treatment. SAE: any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the subject at immediate risk of death; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; any other medically important event that, in the opinion of the Investigator, may jeopardize the subject or may require intervention to prevent one of the other outcomes. An AE was considered treatment-emergent if it occurred after the start of study treatment or was present prior to the start of study treatment but subsequently worsened.
Time Frame: Day 1 up to end of Safety Follow-up (9 weeks)
Population: Safety population: participants who received at least 1 dose of study treatment (BG00012/BG00012 placebo).
Measure: Number; unit: participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 43 | 42
participants
  Any event | 24 | 24 | 26 | 26
  Moderate or severe event | 10 | 13 | 12 | 11
  Severe event | 0 | 4 | 4 | 1
  Related event | 8 | 17 | 16 | 18
  Serious event | 0 | 1 | 0 | 0
  Discontinuation of treatment due to an event | 2 | 4 | 6 | 3
  Withdrawal from study due to an event | 2 | 4 | 6 | 3

18. Secondary Outcome: Clinical Laboratory Shifts From Baseline in Reported Values: Hematology
Description: Number of participants with clinical laboratory shifts from baseline in hematology values. Shift to low includes normal to low, high to low, and unknown to low. Shift to high includes normal to high, low to high, and unknown to high. abs=absolute
Time Frame: Day 1 to Week 8
Population: Safety population: participants who received at least 1 dose of study treatment (BG00012/BG00012 placebo); n=number of participants whose baseline value was not low (or high) and who had at least 1 post-baseline value.
Measure: Number; unit: participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 43 | 42
participants
  White blood cells: shift to low; n=43, 43, 43, 41 | 0 | 2 | 0 | 0
  White blood cells: shift to high; n=44, 43, 43, 42 | 0 | 0 | 1 | 0
  Neutrophils abs: shift to low; n=42, 42, 42, 41 | 3 | 6 | 2 | 2
  Neutrophils abs: shift to high; n=44, 43, 43, 42 | 0 | 0 | 0 | 1
  Lymphocytes abs: shift to low; n=43, 43, 43, 41 | 1 | 5 | 2 | 3
  Lymphocytes abs: shift to high; n=44, 43, 42, 42 | 0 | 0 | 0 | 0
  Monocytes abs: shift to low; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Monocytes abs: shift to high; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Eosinophils abs: shift to low; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Eosinophils abs: shift to high; n=44, 43, 43, 42 | 0 | 5 | 6 | 6
  Basophils abs: shift to high; n=44, 43, 43, 42 | 0 | 1 | 1 | 0
  Red blood cells: shift to low; n=44, 43, 43, 40 | 0 | 2 | 0 | 0
  Red blood cells: shift to high; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Hemoglobin: shift to low; n=43, 41, 43, 42 | 1 | 3 | 1 | 0
  Hemoglobin: shift to high; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Hematocrit: shift to low; n=44, 43, 43, 42 | 0 | 2 | 0 | 0
  Hematocrit: shift to high; n=43, 43, 43, 42 | 0 | 0 | 0 | 1
  Platelets: shift to low; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Platelets: shift to high; n=44, 41, 43, 42 | 0 | 0 | 1 | 1

19. Secondary Outcome: Clinical Laboratory Shifts From Baseline in Reported Values: Blood Chemistry
Description: Number of participants with clinical laboratory shifts from baseline in blood chemistry values. Shift to low includes normal to low, high to low, and unknown to low. Shift to high includes normal to high, low to high, and unknown to high. ALP=alkaline phosphatase, ALT=alanine aminotransferase, AST=aspartate aminotransferase, GGT=gamma-glutamyl transferase, LDH=lactate dehydrogenase, BUN=blood urea nitrogen.
Time Frame: Day 1 to Week 8
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 44 | 43
participants
  ALP: shift to high; n=44, 42, 43, 42 | 0 | 0 | 0 | 0
  ALT: shift to high; n=44, 42, 43, 42 | 1 | 2 | 5 | 2
  AST: shift to high; n=44, 43, 43, 41 | 2 | 3 | 4 | 1
  GGT: shift to high; n=44, 41, 43, 42 | 0 | 0 | 2 | 0
  LDH: shift to low; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  LDH: shift to high; n=44, 43, 43, 42 | 0 | 0 | 1 | 0
  Total bilirubin: shift to high; n=44, 42, 42, 40 | 1 | 1 | 0 | 1
  BUN: shift to low; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  BUN: shift to high; n=44, 43, 41, 42 | 1 | 0 | 1 | 1
  Creatinine: shift to low; n=44, 43, 43, 42 | 0 | 1 | 0 | 0
  Creatinine: shift to high; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Uric Acid: shift to low; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Uric Acid: shift to high; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Sodium: shift to low; n=44, 43, 43, 42 | 1 | 0 | 0 | 0
  Sodium: shift to high; n=44, 43, 43, 42 | 0 | 0 | 1 | 0
  Potassium: shift to low: n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Potassium: shift to high: n=44, 42, 42, 41 | 1 | 1 | 1 | 0
  Chloride: shift to low; n=44, 43, 43, 42 | 1 | 0 | 0 | 0
  Chloride: shift to high; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Bicarbonate: shift to low; n=44, 43, 43, 42 | 1 | 1 | 1 | 0
  Bicarbonate: shift to high; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Calcium: shift to low; n=44, 42, 43, 42 | 0 | 0 | 1 | 0
  Calcium: shift to high; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Glucose: shift to low; n=43, 43, 41, 41 | 3 | 1 | 1 | 2
  Glucose: shift to high; n=44, 43, 43, 42 | 1 | 0 | 0 | 0
  Magnesium: shift to low; n=44, 43, 43, 42 | 1 | 0 | 0 | 1
  Magnesium: shift to high; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Phosphorus: shift to low; n=44, 43, 43, 41 | 0 | 1 | 0 | 0
  Phosphorus: shift to high; n=44, 43, 43, 42 | 0 | 0 | 0 | 1
  Albumin: shift to low; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Albumin: shift to high; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Direct bilirubin: shift to high; n=44, 43, 43, 40 | 0 | 0 | 0 | 0
  Total protein: shift to low; n=44, 41, 43, 41 | 0 | 0 | 1 | 0
  Total protein: shift to high; n=44, 43, 43, 42 | 0 | 0 | 0 | 0

20. Secondary Outcome: Clinical Laboratory Shifts From Baseline in Reported Values: Urinalysis
Description: Number of participants with clinical laboratory shifts from baseline in urinalysis values.Shift to low includes normal to low, high to low, and unknown to low. Shift to high includes normal to high, low to high, and unknown to high. Shift to positive includes negative to positive and unknown to positive. RBC=red blood cells, WBC=white blood cells.
Time Frame: Day 1 to Week 8
Population: Safety population: participants who received at least 1 dose of study treatment (BG00012/BG00012 placebo); n=number of participants whose baseline value was not low (or high or positive) and who had at least 1 post-baseline value.
Measure: Number; unit: participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 43 | 42
participants
  Specific gravity: shift to low; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Specific gravity: shift to high; n=44, 42, 43, 42 | 0 | 0 | 2 | 0
  pH: shift to low; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  pH: shift to high; n=44, 43, 43, 42 | 0 | 0 | 0 | 0
  Blood: shift to positive; n=42, 39, 39, 42 | 3 | 6 | 1 | 2
  Color: shift to positive; n=41, 43, 41, 39 | 2 | 1 | 4 | 5
  Glucose: shift to positive; n=44, 43, 43, 41 | 0 | 2 | 1 | 0
  Ketones: shift to positive; n=44, 43, 43, 42 | 1 | 7 | 9 | 6
  Protein: shift to positive; n=44, 41, 43, 41 | 0 | 1 | 1 | 1
  Microscopic RBC; n=44, 40, 40, 41 | 3 | 4 | 1 | 2
  Microscopic WBC; n=43, 40, 41, 42 | 4 | 9 | 3 | 3

21. Secondary Outcome: Number of Participants With Abnormalities in Vital Signs
Description: ↑=increase; ↓=decrease; BL=baseline; bpm=beats per minute; SBP=systolic blood pressure; DBP=diastolic blood pressure; b/m=breaths per minute
Time Frame: Day 1 to Week 8
Population: Safety population: participants who received at least 1 dose of study treatment (BG00012/BG00012 placebo); n=number of participants who had a baseline value and had at least 1 post-baseline value.
Measure: Number; unit: participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 43 | 42
participants
  Temperature >38°C + ↑ from BL of ≥1°C | 0 | 0 | 0 | 0
  Pulse >120 bpm or ↑ from BL of >20 bpm | 8 | 10 | 20 | 17
  Pulse <50 bpm or ↓ from BL of >20 bpm | 11 | 4 | 3 | 4
  SBP >180 mm Hg or ↑ from BL of >40 mm Hg | 1 | 0 | 0 | 0
  SBP <90 mm Hg or ↓ from BL of >30 mm Hg | 1 | 2 | 1 | 1
  DBP >105 mm Hg or ↑ from BL of >30 mm Hg | 0 | 0 | 0 | 0
  DBP <50 mm Hg or ↓ from BL of >20 mm Hg | 1 | 3 | 0 | 1
  Respiration rate >25 b/m or ↑ from BL of ≥50% | 1 | 2 | 3 | 3
  Respiration rate 10 b/m or ↓ from BL of ≥50% | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Shifts From Baseline in Electrocardiogram (ECG) Results
Description: Shift to 'abnormal, not adverse event' includes unknown or normal to 'abnormal, not adverse event.' Shift to 'abnormal, adverse event' includes unknown or normal to 'abnormal, adverse event.'
Time Frame: Day 1 to Week 8
Population: Safety population: participants who received at least 1 dose of study treatment (BG00012/BG00012 placebo); n=number of participants whose baseline value was not abnormal and who had at least 1 post-baseline value.
Measure: Number; unit: participants
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 43 | 42
participants
  Shift to abnormal, not adverse event | 2 | 3 | 2 | 4
  Shift to abnormal, adverse event | 0 | 0 | 0 | 0

23. Secondary Outcome: Duration of Flushing Events During the Overall Treatment Period, Based on MFSS
Description: For participants with more than 1 flushing episode during a visit interval, the average duration for the visit interval was used. The average duration is calculated as: the total duration of all flushing episodes / the total number of flushing episodes.
Time Frame: Day 1 to Week 8
Population: Participants with a flushing event.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 18 | 39 | 35 | 41
minutes | 98.4 (92.04) | 63.2 (34.55) | 69.8 (78.09) | 68.9 (52.82)
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Test type: Superiority or Other; Mean Difference (Final Values) = 6.6, 95% CI 2-sided [-20.9 to 34.1], Standard Error of Mean 13.79 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Test type: Superiority or Other; Mean Difference (Final Values) = 5.8, 95% CI 2-sided [-14.2 to 25.7], Standard Error of Mean 10.03 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

24. Secondary Outcome: Duration of Flushing Events During the Weeks 1 to 4 (Combined), Based on MFSS
Description: as for outcome 23
Time Frame: Week 1 to Week 4
Population: Participants with a flushing event.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 18 | 37 | 31 | 41
minutes | 117.6 (143.90) | 67.6 (43.83) | 89.8 (140.67) | 69.2 (53.00)
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Test type: Superiority or Other; Mean Difference (Final Values) = 22.2, 95% CI 2-sided [-26.5 to 70.9], Standard Error of Mean 24.40 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Test type: Superiority or Other; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-20.5 to 23.6], Standard Error of Mean 11.08 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

25. Secondary Outcome: Duration of Flushing Events During the Weeks 5 to 8 (Combined), Based on MFSS
Description: as for outcome 23
Time Frame: Week 5 to Week 8
Population: Participants with a flushing event.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 10 | 32 | 26 | 28
minutes | 113.2 (160.82) | 55.7 (32.37) | 73.2 (66.34) | 56.0 (35.79)
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Test type: Superiority or Other; Mean Difference (Final Values) = 17.5, 95% CI 2-sided [-9.2 to 44.2], Standard Error of Mean 13.32 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Test type: Superiority or Other; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-17.2 to 18.0], Standard Error of Mean 8.80 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

26. Secondary Outcome: Duration of Acute GI Episodes During the Overall Treatment Period, Based on MAGISS
Description: Duration is calculated as follows: [(GI side effect) end date/time - (GI side effect) start date/time]/3600. For GI side effects with no end date, the end date is imputed using the last diary date/time. For subjects with more than 1 GI episode during a visit interval, the average duration for the study visit interval is used. The average duration is calculated as the total duration of the GI side effect / the total number of GI side effects.
Time Frame: Day 1 to Week 8
Population: Participants in the safety population who have at least 1 diary entry of the relevant questionnaire data during the visit interval; n=number of participants with the given GI episode during the visit interval.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 43 | 42
hours
  Nausea; n=12, 21, 21, 22 | 9.74 (17.008) | 7.05 (10.498) | 10.01 (18.283) | 2.98 (3.247)
  Diarrhea; n=20, 20 17, 15 | 5.57 (10.037) | 2.92 (3.329) | 14.66 (32.686) | 4.97 (9.687)
  Upper abdominal pain; n=17, 14, 19, 19 | 19.08 (46.873) | 6.67 (16.916) | 15.88 (25.307) | 3.83 (5.712)
  Lower abdominal pain; n=12, 19, 17, 16 | 6.65 (5.307) | 13.93 (26.850) | 10.84 (16.312) | 7.75 (10.456)
  Vomiting; n=3, 3, 3, 2 | 5.87 (5.033) | 10.08 (8.755) | 1.88 (2.717) | 0.75 (0.707)
  Indigestion; n=12, 13, 12, 12 | 4.76 (8.203) | 16.49 (28.865) | 3.80 (2.543) | 4.91 (8.263)
  Constipation; n=6, 8, 13, 11 | 20.49 (12.040) | 28.20 (35.425) | 14.26 (9.783) | 20.90 (18.060)
  Bloating; n=14, 14, 21, 12 | 9.50 (9.066) | 16.91 (27.128) | 9.68 (10.108) | 77.24 (125.961)
  Flatulence; n=23, 20, 22, 20 | 16.41 (44.149) | 9.06 (9.626) | 68.93 (290.248) | 63.84 (180.597)
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Nausea; Test type: Superiority or Other; Mean Difference (Final Values) = 2.96, 95% CI 2-sided [-6.34 to 12.26], Standard Error of Mean 4.601 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Nausea; Test type: Superiority or Other; Mean Difference (Final Values) = -4.07, 95% CI 2-sided [-8.81 to 0.67], Standard Error of Mean 2.347 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 3: Comparison: BG00012 vs BG00012 + ASA; Diarrhea; Test type: Superiority or Other; Mean Difference (Final Values) = 11.74, 95% CI 2-sided [-3.15 to 26.63], Standard Error of Mean 7.335 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 4: Comparison: BG00012 vs BG00012 Slow Titration; Diarrhea; Test type: Superiority or Other; Mean Difference (Final Values) = 2.05, 95% CI 2-sided [-2.67 to 6.77], Standard Error of Mean 2.321 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 5: Comparison: BG00012 vs BG00012 + ASA; Upper abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = 9.21, 95% CI 2-sided [-6.72 to 25.14], Standard Error of Mean 7.812 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 6: Comparison: BG00012 vs BG00012 Slow Titration; Upper abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = -2.84, 95% CI 2-sided [-11.31 to 5.63], Standard Error of Mean 4.152 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 7: Comparison: BG00012 vs BG00012 + ASA; Lower abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = -3.09, 95% CI 2-sided [-18.36 to 12.19], Standard Error of Mean 7.516 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 8: Comparison: BG00012 vs BG00012 Slow Titration; Lower abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = -6.18, 95% CI 2-sided [-20.71 to 8.35], Standard Error of Mean 7.141 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 9: Comparison: BG00012 vs BG00012 + ASA; Vomiting; Test type: Superiority or Other; Mean Difference (Final Values) = -8.21, 95% CI 2-sided [-22.90 to 6.49], Standard Error of Mean 5.292 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 10: Comparison: BG00012 vs BG00012 Slow Titration; Vomiting; Test type: Superiority or Other; Mean Difference (Final Values) = -9.33, 95% CI 2-sided [-30.13 to 11.47], Standard Error of Mean 6.536 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 11: Comparison: BG00012 vs BG00012 + ASA; Indigestion; Test type: Superiority or Other; Mean Difference (Final Values) = -12.69, 95% CI 2-sided [-30.02 to 4.63], Standard Error of Mean 8.376 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 12: Comparison: BG00012 vs BG00012 Slow Titration; Indigestion; Test type: Superiority or Other; Mean Difference (Final Values) = -11.58, 95% CI 2-sided [-29.48 to 6.32], Standard Error of Mean 8.654 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 13: Comparison: BG00012 vs BG00012 + ASA; Constipation; Test type: Superiority or Other; Mean Difference (Final Values) = -13.93, 95% CI 2-sided [-35.44 to 7.57], Standard Error of Mean 10.274 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 14: Comparison: BG00012 vs BG00012 Slow Titration; Constipation; Test type: Superiority or Other; Mean Difference (Final Values) = -7.29, 95% CI 2-sided [-33.39 to 18.81], Standard Error of Mean 12.369 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 15: Comparison: BG00012 vs BG00012 + ASA; Bloating; Test type: Superiority or Other; Mean Difference (Final Values) = -7.24, 95% CI 2-sided [-20.40 to 5.93], Standard Error of Mean 6.472 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 16: Comparison: BG00012 vs BG00012 Slow Titration; Bloating; Test type: Superiority or Other; Mean Difference (Final Values) = 60.33, 95% CI 2-sided [-10.78 to 131.4], Standard Error of Mean 34.455 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 17: Comparison: BG00012 vs BG00012 + ASA; Flatulence; Test type: Superiority or Other; Mean Difference (Final Values) = 59.87, 95% CI 2-sided [-71.51 to 191.2], Standard Error of Mean 65.007 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 18: Comparison: BG00012 vs BG00012 Slow Titration; Flatulence; Test type: Superiority or Other; Mean Difference (Final Values) = 54.78, 95% CI 2-sided [-27.09 to 136.6], Standard Error of Mean 40.440 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

27. Secondary Outcome: Duration of Acute GI Episodes During Weeks 1 to 4 (Combined), Based on MAGISS
Description: as for outcome 26
Time Frame: Week 1 to Week 4
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 43 | 42
hours
  Nausea; n=10, 18, 18, 20 | 10.47 (18.678) | 7.23 (10.916) | 11.18 (19.568) | 2.86 (3.359)
  Diarrhea; n=13, 20, 14, 14 | 5.20 (11.309) | 2.53 (3.013) | 16.04 (35.945) | 4.97 (10.074)
  Upper abdominal pain; n=14, 14, 17, 15 | 21.37 (51.620) | 6.81 (16.876) | 17.65 (26.294) | 4.31 (6.350)
  Lower abdominal pain; n=9, 18, 14, 13 | 5.40 (4.658) | 14.20 (27.637) | 12.51 (17.621) | 6.30 (6.080)
  Vomiting; n=2, 2, 2, 2 | 4.31 (5.999) | 5.63 (5.834) | 2.53 (3.500) | 0.75 (0.707)
  Indigestion; n=11, 11, 9, 11 | 5.08 (8.552) | 29.00 (48.416) | 3.93 (2.873) | 5.05 (8.665)
  Constipation; n=4, 8, 11, 11 | 17.05 (7.452) | 27.61 (35.177) | 15.12 (7.761) | 21.28 (19.298)
  Bloating; n=9, 14, 19, 11 | 6.70 (6.792) | 13.81 (25.321) | 11.07 (10.631) | 95.69 (186.884)
  Flatulence; n=21, 17, 22, 19 | 12.83 (27.948) | 9.34 (12.946) | 35.86 (134.748) | 61.13 (168.572)
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Nausea; Test type: Superiority or Other; Mean Difference (Final Values) = 3.95, 95% CI 2-sided [-6.79 to 14.68], Standard Error of Mean 5.281 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Nausea; Test type: Superiority or Other; Mean Difference (Final Values) = -4.37, 95% CI 2-sided [-9.57 to 0.83], Standard Error of Mean 2.563 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 3: Comparison: BG00012 vs BG00012 + ASA; Diarrhea; Test type: Superiority or Other; Mean Difference (Final Values) = 13.51, 95% CI 2-sided [-2.84 to 29.86], Standard Error of Mean 8.024 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 4: Comparison: BG00012 vs BG00012 Slow Titration; Diarrhea; Test type: Superiority or Other; Mean Difference (Final Values) = 2.44, 95% CI 2-sided [-2.41 to 7.29], Standard Error of Mean 2.379 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 5: Comparison: BG00012 vs BG00012 + ASA; Upper abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = 10.84, 95% CI 2-sided [-5.81 to 27.50], Standard Error of Mean 8.143 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 6: Comparison: BG00012 vs BG00012 Slow Titration; Upper abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = -2.50, 95% CI 2-sided [-12.08 to 7.09], Standard Error of Mean 4.671 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 7: Comparison: BG00012 vs BG00012 + ASA; Lower abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = -1.69, 95% CI 2-sided [-19.03 to 15.64], Standard Error of Mean 8.488 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 8: Comparison: BG00012 vs BG00012 Slow Titration; Lower abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = -7.91, 95% CI 2-sided [-23.93 to 8.11], Standard Error of Mean 7.832 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 9: Comparison: BG00012 vs BG00012 + ASA; Vomiting; Test type: Superiority or Other; Mean Difference (Final Values) = -3.10, 95% CI 2-sided [-23.80 to 17.60], Standard Error of Mean 4.811 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 10: Comparison: BG00012 vs BG00012 Slow Titration; Vomiting; Test type: Superiority or Other; Mean Difference (Final Values) = -4.88, 95% CI 2-sided [-22.75 to 13.00], Standard Error of Mean 4.155 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 11: Comparison: BG00012 vs BG00012 + ASA; Indigestion; Test type: Superiority or Other; Mean Difference (Final Values) = -25.08, 95% CI 2-sided [-59.20 to 9.05], Standard Error of Mean 16.243 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 12: Comparison: BG00012 vs BG00012 Slow Titration; Indigestion; Test type: Superiority or Other; Mean Difference (Final Values) = -23.95, 95% CI 2-sided [-54.89 to 6.98], Standard Error of Mean 14.830 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 13: Comparison: BG00012 vs BG00012 + ASA; Constipation; Test type: Superiority or Other; Mean Difference (Final Values) = -12.49, 95% CI 2-sided [-35.38 to 10.39], Standard Error of Mean 10.847 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 14: Comparison: BG00012 vs BG00012 Slow Titration; Constipation; Test type: Superiority or Other; Mean Difference (Final Values) = -6.33, 95% CI 2-sided [-32.79 to 20.13], Standard Error of Mean 12.542 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 15: Comparison: BG00012 vs BG00012 + ASA; Bloating; Test type: Superiority or Other; Mean Difference (Final Values) = -2.73, 95% CI 2-sided [-15.87 to 10.41], Standard Error of Mean 6.442 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 16: Comparison: BG00012 vs BG00012 Slow Titration; Bloating; Test type: Superiority or Other; Mean Difference (Final Values) = 81.89, 95% CI 2-sided [-22.04 to 185.8], Standard Error of Mean 50.239 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 17: Comparison: BG00012 vs BG00012 + ASA; Flatulence; Test type: Superiority or Other; Mean Difference (Final Values) = 26.52, 95% CI 2-sided [-40.13 to 93.18], Standard Error of Mean 32.896 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 18: Comparison: BG00012 vs BG00012 Slow Titration; Flatulence; Test type: Superiority or Other; Mean Difference (Final Values) = 51.78, 95% CI 2-sided [-31.65 to 135.2], Standard Error of Mean 41.055 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

28. Secondary Outcome: Duration of Acute GI Episodes During Weeks 5 to 8 (Combined), Based on MAGISS
Description: as for outcome 26
Time Frame: Week 5 to Week 8
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Number analyzed (Participants) | 44 | 43 | 43 | 42
hours
  Nausea; n=4, 9, 6, 9 | 3.96 (3.668) | 4.34 (6.256) | 2.66 (1.390) | 2.34 (1.904)
  Diarrhea; n=12, 13, 6, 8 | 4.50 (6.389) | 6.62 (12.782) | 7.05 (8.002) | 2.14 (2.007)
  Upper abdominal pain; n=6, 5, 5, 5 | 5.29 (5.785) | 1.12 (0.965) | 1.86 (1.491) | 1.73 (1.440)
  Lower abdominal pain; n=7, 5, 5, 9 | 6.63 (7.739) | 3.98 (3.516) | 2.84 (1.477) | 22.54 (61.180)
  Vomiting; n=1, 1, 1, 0 | 9.00 (NA) — n=1 participant | 19.00 (NA) — n=1 participant | 0.58 (NA) — n=1 participant | NA (NA) — n=0 participants
  Indigestion; n=6, 7, 7, 5 | 2.43 (1.569) | 2.57 (2.586) | 5.02 (6.944) | 1.63 (1.101)
  Constipation; n=5, 2, 4, 4 | 23.35 (17.110) | 15.47 (21.143) | 21.30 (23.181) | 18.24 (8.644)
  Bloating; n=7, 8, 7, 8 | 12.49 (10.595) | 18.52 (25.682) | 4.16 (3.018) | 85.64 (115.872)
  Flatulence; n=9, 13, 7, 10 | 44.67 (112.426) | 7.21 (10.051) | 105.86 (275.125) | 18.48 (26.347)
Statistical Analysis 1: Comparison: BG00012 vs BG00012 + ASA; Nausea; Test type: Superiority or Other; Mean Difference (Final Values) = -1.68, 95% CI 2-sided [-7.35 to 3.99], Standard Error of Mean 2.626 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 2: Comparison: BG00012 vs BG00012 Slow Titration; Nausea; Test type: Superiority or Other; Mean Difference (Final Values) = -2.00, 95% CI 2-sided [-6.62 to 2.62], Standard Error of Mean 2.180 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 3: Comparison: BG00012 vs BG00012 + ASA; Diarrhea; Test type: Superiority or Other; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-11.64 to 12.49], Standard Error of Mean 5.717 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 4: Comparison: BG00012 vs BG00012 Slow Titration; Diarrhea; Test type: Superiority or Other; Mean Difference (Final Values) = -4.48, 95% CI 2-sided [-14.11 to 5.14], Standard Error of Mean 4.597
Statistical Analysis 5: Comparison: BG00012 vs BG00012 + ASA; Upper abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [-1.10 to 2.57], Standard Error of Mean 0.794 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 6: Comparison: BG00012 vs BG00012 Slow Titration; Upper abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-1.17 to 2.40], Standard Error of Mean 0.775 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 7: Comparison: BG00012 vs BG00012 + ASA; Lower abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = -1.14, 95% CI 2-sided [-5.08 to 2.79], Standard Error of Mean 1.705 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 8: Comparison: BG00012 vs BG00012 Slow Titration; Lower abdominal pain; Test type: Superiority or Other; Mean Difference (Final Values) = 18.56, 95% CI 2-sided [-42.19 to 79.32], Standard Error of Mean 27.886 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 9: Comparison: BG00012 vs BG00012 + ASA; Indigestion; Test type: Superiority or Other; Mean Difference (Final Values) = 2.46, 95% CI 2-sided [-3.65 to 8.56], Standard Error of Mean 2.801 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 10: Comparison: BG00012 vs BG00012 Slow Titration; Indigestion; Test type: Superiority or Other; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-3.71 to 1.83], Standard Error of Mean 1.242 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 11: Comparison: BG00012 vs BG00012 + ASA; Constipation; Test type: Superiority or Other; Mean Difference (Final Values) = 5.83, 95% CI 2-sided [-48.73 to 60.38], Standard Error of Mean 19.649 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 12: Comparison: BG00012 vs BG00012 Slow Titration; Constipation; Test type: Superiority or Other; Mean Difference (Final Values) = 2.76, 95% CI 2-sided [-28.38 to 33.91], Standard Error of Mean 11.219 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 13: Comparison: BG00012 vs BG00012 + ASA; Bloating; Test type: Superiority or Other; Mean Difference (Final Values) = -14.36, 95% CI 2-sided [-35.56 to 6.83], Standard Error of Mean 9.811 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 14: Comparison: BG00012 vs BG00012 Slow Titration; Bloating; Test type: Superiority or Other; Mean Difference (Final Values) = 67.12, 95% CI 2-sided [-22.88 to 157.1], Standard Error of Mean 41.961 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 15: Comparison: BG00012 vs BG00012 + ASA; Flatulence; Test type: Superiority or Other; Mean Difference (Final Values) = 98.65, 95% CI 2-sided [-58.01 to 255.3], Standard Error of Mean 74.566 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect
Statistical Analysis 16: Comparison: BG00012 vs BG00012 Slow Titration; Flatulence; Test type: Superiority or Other; Mean Difference (Final Values) = 11.27, 95% CI 2-sided [-5.22 to 27.76], Standard Error of Mean 7.928 — Reference arm is BG00012 240 mg BID; negative values means reduced side effect

ADVERSE EVENTS:
Time Frame: AEs: from the administration of the first dose of study treatment to the Safety Follow-up (approximately 9 weeks). SAEs: from signing of informed consent to the Safety Follow-up (up to approximately 13 weeks).
Description: Flushing and GI events/symptoms captured separately in the eDiary were not recorded on the AE eCRF unless the events/symptoms led to discontinuation or withdrawal from the study, were classified as SAEs, or were ongoing at the final eDiary entry.
Arm/Group | Placebo | BG00012 | BG00012 + ASA | BG00012 Slow Titration
Serious Adverse Events (participants affected / at risk) | 0/44 | 1/43 | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 5/44 | 12/43 | 15/43 | 12/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=44) | BG00012 (N=43) | BG00012 + ASA (N=43) | BG00012 Slow Titration (N=42)
Ovarian germ cell teratoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=44) | BG00012 (N=43) | BG00012 + ASA (N=43) | BG00012 Slow Titration (N=42)
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 7 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 2
Headache (Nervous system disorders) | 4 | 9 | 2 | 9
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 5 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.